CLINICAL TRIAL: NCT07330622
Title: Polish Registry of Percutaneous Coronary Intervention for Chronic Total Occlusions (POL-CTO Registry)
Brief Title: Polish Registry of Percutaneous Coronary Intervention for Chronic Total Occlusions
Acronym: POL-CTO
Status: Recruiting | Type: Observational
Sponsor: National Institute of Cardiology, Warsaw, Poland (Other)
Collaborators: Polish Cardiac Society (Other)
Responsible Party: Sponsor
Other Study IDs: 4.49/III/24
Record Dates: First submitted 2025-12-29; First posted 2026-01-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-10

CONDITIONS: Coronary Occlusion; Percutaneous Coronary Intervention
Keywords: coronary artery disease; percutaneous coronary intervention; coronary chronic total occlusion
MeSH Terms: conditions — Coronary Occlusion; Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to evaluate the safety, efficacy, and clinical outcomes of percutaneous coronary intervention (PCI) for chronic total occlusions (CTO) in patients treated in contemporary clinical practice in Poland.

The main questions it aims to answer are:

* What are the rates of procedural success and periprocedural complications of CTO PCI in routine clinical practice?
* How do CTO PCI strategies and techniques, intravascular imaging, different treatment strategies, and mechanical circulatory support affect clinical outcomes?
* How do clinical outcomes differ among different patient subgroups?
* Can artificial intelligence-based analysis predict clinical and quality-of-life outcomes after CTO PCI?

Patients undergoing CTO PCI as part of their standard medical care will be prospectively enrolled in a national, multicenter registry, with clinical, procedural, and follow-up data collected to evaluate real-world outcomes.

DETAILED DESCRIPTION:
Coronary chronic total occlusions (CTO) are diagnosed in approximately 20% of patients undergoing invasive coronary angiography, and their presence is associated with significantly reduced quality of life and worse long-term prognosis compared with patients without a CTO. Successful CTO recanalization improves quality of life, regional and global left ventricular function, and reduces myocardial ischemia in most patients. Over the past decade, the success rate of percutaneous coronary intervention (PCI) for CTO has increased substantially, largely due to advances in dedicated equipment and specialized procedural techniques. Concurrently, there is a growing need to evaluate the safety and effectiveness of contemporary CTO PCI techniques in selected patient populations.

The aim of the POL-CTO registry is to expand current knowledge regarding the safety and efficacy of CTO PCI in the contemporary Polish population across a broad range of clinical scenarios. Specifically, the registry will examine the incidence and management of periprocedural complications, as well as the impact of post-procedural cardiac injury markers on clinical outcomes. Comparative analyses of PCI performed with versus without intravascular imaging, along with different treatment strategies (drug-coated balloon [DCB], drug-eluting stent [DES], or hybrid approaches), will be conducted. Additional objectives include evaluating the safety of PCI with mechanical circulatory support and predicting quality-of-life improvement using artificial intelligence-based analysis of baseline electrocardiograms. Finally, the study will focus on CTO PCI outcomes in high-risk subgroups, including patients with low ejection fraction, frailty syndrome, severe coronary calcification, diabetes, prior transcatheter aortic valve implantation, prior coronary artery bypass grafting, and in-stent CTO.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing CTO PCI based on clinical grounds

Exclusion Criteria:

* Age <18 years
* Patient's refusal to participate in the registry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients undergoing CTO PCI at participating centers.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2025-05-21 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Technical success | procedural (1 day)
  Achievement of Thrombolysis In Myocardial Infarction grade 3 flow in all ≥2.5-mm distal branches with <30% residual stenosis.

SECONDARY OUTCOMES:
Total procedure time | procedural (1 day)
  Total procedure time in minutes.
Fluoroscopy time | procedural (1 day)
  Fluoroscopy time in minutes.
Radiation dose | procedural (1 day)
  Total radiation dose in Gy and uGycm2.
Contrast volume | procedural (1 day)
  Total contrast volume in mL.
Number and type of procedural complications | procedural (1 day)
  Total number and specification of procedural complications (death, non-fatal myocardial infarction, cardiac tamponade requiring pericardiocentesis, coronary perforation, stroke, major bleeding according to Bleeding Academic Research Consortium).
Successful guidewire crossing through CTO | procedural (1 day)
  Rate of successful guidewire crossing through CTO.
Time of successful guidewire crossing | procedural (1 day)
  Time of successful guidewire crossing through CTO in minutes defined as the time from starting primary CTO PCI strategy to the time of successful CTO recanalization using any technique.
Target lesion failure | in-hospital (2-5 days)
  Total number of cardiac death, target vessel-related myocardial infarction or clinically-driven target lesion revascularization
Target lesion failure | 1 year
  otal number of cardiac death, target vessel-related myocardial infarction or clinically-driven target lesion revascularization
Death | 1 year
  Any death

CONTACTS AND LOCATIONS:
Locations (21):
- Poland (21):
  - Medical University of Białystok, Bialystok
  - Szpital Zachodni, Grodzisk Mazowiecki
  - Specialist Hospital in Inowrocław, Inowrocław
  - Medical University of Silesia, Katowice
  - Institute of Cardiology, Krakow
  - St. John Paul II Hospital, Krakow
  - Copper Health Centre Inc., Lubin
  - 1st Military Clinical Hospital, Lublin
  - Hospital of the Ministry of the Interior and Administration, Lublin
  - University of Applied Science in Nowy Sącz, Nowy Sącz
  - Masovian Specialist Hospital, Ostrołęka
  - Poznań University of Medical Sciences, Poznan
  - Samodzielny Publiczny Zakład Opieki Zdrowotnej w Puławach, Puławy
  - Specialistic Hospital, Radom
  - The Ministry of Internal Affairs and Administration Hospital, Rzeszów
  - Military Institute of Medicine - National Research Institute, Warsaw
  - National Institute of Cardiology, Warsaw
  - The Doctor Sokolowski Hospital, Wałbrzych
  - Military Hospital in Wrocław, Wroclaw
  - University Hospital in Wroclaw, Wroclaw
  - Provincial Hospital in Łomża, Łomża